CLINICAL TRIAL: NCT01849211
Title: Influence of a Neuromuscular Block on Face Mask Ventilation Conditions During Induction of Anaesthesia
Brief Title: Influence of Neuromuscular Block on Mask Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kreiskrankenhaus Dormagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: diffmask
Record Dates: First submitted 2013-04-25; First posted 2013-05-08 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2018-03

CONDITIONS: Effect of a Neuromuscular Block on Ventilation
Keywords: ventilation; face mask; NMBA
MeSH Terms: conditions — Respiratory Aspiration | interventions — Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neuromuscular block (Other)
  Interventions: Drug: rocuronium

INTERVENTIONS:
Drug: rocuronium

SUMMARY:
Difficult mask ventilation might lead to a life-threatening situation, if endotracheal intubation is also impossible and neuromuscular blocking agents (NMBA) inhibit spontaneous ventilation. However, controversies exist if NMBA improve or impede face mask ventilation. Therefore, the effect of NMBAs on mask ventilation is assessed in patients with predictors for difficult face mask ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with risk factors for difficult face mask ventilation
* Patients scheduled for general anaesthesia with endotracheal intubation

Exclusion Criteria:

* Increased Risk for pulmonary aspiration
* scheduled for awake fiberoptic intubation
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2017-04 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
minute volume | 15 min (from Induction of anaesthesia until onset of NMBA )

SECONDARY OUTCOMES:
incidence of difficult mask ventilation - tidal volume < 150 ml | 15 min

OTHER OUTCOMES:
airway pressure | 15 min
  measurement of peak airway pressure

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Soltesz, MD, Principal Investigator — KKH Dormagen
Locations (1):
- KKH Dormagen, Dormagen, Germany